CLINICAL TRIAL: NCT01688011
Title: Connect® Myeloid: The Myelofibrosis (MF), Myelodysplastic Syndromes (MDS) and Acute Myeloid Leukemia (AML) Disease Registry
Brief Title: Connect® Myeloid Disease Registry
Status: Terminated | Type: Observational
Why Stopped: Business objectives have changed
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Other Study IDs: AZA-MDS-006; Connect® MDS/AML Registry (Other: BMS)
Record Dates: First submitted 2012-09-14; First posted 2012-09-19 (Estimated); Last update posted 2025-07-03 (Actual); Status verified 2025-06

CONDITIONS: Primary Myelofibrosis; Myelodysplastic Syndromes; Leukemia, Myeloid, Acute
Keywords: Myelodysplastic syndromes; MDS; Acute myeloid leukemia; AML; Registry; Connect®; ICUS; Idiopathic Cytopenias of Undetermined Significance; Myelofibrosis; MF; Myelodysplastic/Myeloproliferative overlap syndromes; MDS/MPN overlap syndromes
MeSH Terms: conditions — Primary Myelofibrosis; Myelodysplastic Syndromes; Leukemia, Myeloid, Acute | interventions — luspatercept

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 8 Years
Biospecimen Retention: Samples With DNA — Perform molecular and cellular correlative studies on blood/bone marrow and oral epithelial cell samples.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (7):
- Newly diagnosed Lower-Risk Myelodysplastic Syndromes (LR-MDS): Newly diagnosed lower risk MDS patients as determined by International Prognostic Scoring System (IPSS).
- Newly diagnosed Higher-Risk Myelodysplastic Syndromes (HR-MDS): Newly diagnosed higher risk MDS patients as determined by International Prognostic Scoring System (IPSS).
- Newly diagnosed Acute Myeloid Leukemia (AML): Newly diagnosed AML patients (≥55 years old, excluding patients with acute promyelocytic leukemia (APL).
- Treated Myelofibrosis (MF): Newly treated MF patients receiving treatment for MF or MF-related cytopenias. This cohort also includes patients with myelodysplastic syndrome (MDS)/myeloproliferative neoplasm (MPN) overlap syndromes, excluding juvenile myelomonocytic leukemia (JMML).
- Newly diagnosed Idiopathic cytopenia of undetermined significance (ICUS): Newly diagnosed ICUS patients.
- Treated Lower-Risk Myelodysplastic Syndromes (LR-MDS): Treated LR-MDS patients receiving first active treatment regimen containing at least one non-ESA therapy
- Luspatercept treated cohort (LTC): Participants that have initiated luspatercept treatment for a myeloid malignancy.
  Interventions: Drug: Luspatercept

INTERVENTIONS:
Drug: Luspatercept — Prescribed by treating physician as per product label.
  Groups: Luspatercept treated cohort (LTC)

SUMMARY:
The purpose of the Connect® Myeloid disease registry is to provide unique insights into treatment decisions and treatment patterns as they relate to clinical outcomes of patients with myeloid diseases in routine clinical practice. This disease registry will also evaluate molecular and cellular markers that may provide further prognostic classification which may or may not be predictive of therapy and clinical outcomes.

DETAILED DESCRIPTION:
This Disease Registry will collect data on patient characteristics, treatment patterns and clinical outcomes. The objective is to describe how patients with myeloid diseases are treated; and to build a knowledge base regarding the effectiveness and safety of first line and subsequent treatment regimens in both community and academic settings. Enrolled patients will receive treatment and evaluations for their disease according to the standard of care and routine clinical practice at each study site. All treatments that patients receive for their disease will be recorded, including initial treatment and any subsequent therapy. Data on treatment outcomes, including response rates as measured by the treating physician, evidence of progression, survival, and patient-reported outcomes will be collected quarterly on the electronic CRF.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be able to provide written informed consent form (ICF)
* Must be willing and able to complete baseline and follow-up HRQoL instruments, for which patients must be proficient in either English or Spanish
* AML patients must be at least 55 years of age at the time of informed consent.
* MF, ICUS, and MDS patients must be at least 18 years of age at the time of informed consent.

Newly diagnosed Idiopathic Cytopenias of Undetermined Significance (ICUS), Myelodysplastic Syndromes (MDS), Acute Myeloid Leukemia (AML) patients:

* Newly diagnosed primary or secondary disease. To be considered "newly diagnosed", a patient's confirmed diagnosis must be made no more than 60 days prior to the date of consent signature. (An additional 5-day window [i.e., up to 65 days prior to the date of ICF signature] may be allowed in special circumstance upon sponsor approval)
* Cohort assignment confirmed by central eligibility review. Cohort assignment must also be confirmed by the site.

Myelofibrosis (MF) patients:

* Patients who initiated their first active systemic treatment for MF and/or MF-related cytopenias within 90 days prior to the date of consent signature. This cohort allows the enrollment of subjects with a diagnosis of Myelodysplastic/Myeloproliferative overlap syndromes (MDS/MPN overlap syndrome).
* Cohort assignment is confirmed by the site. Central eligibility review is not required.

Treated Lower-Risk Myelodysplastic Syndromes (LR-MDS) patients:

* Patients who have initiated first active treatment regimen containing at least one non-ESA therapy, within 90 days prior to ICF
* Cohort assignment is confirmed by site. Central eligibility review is not required.

Luspatercept treated patients:

* Patient must have been at least 18 years of age at the start of luspatercept.
* Among LR-MDS patients, patient must have initiated luspatercept on or after September 1, 2023, must be ESA-naïve and luspatercept must be the first active treatment (as monotherapy or part of a treatment regimen) for their disease.
* Among all other myeloid malignancies, there is no date restriction for initiation of luspatercept .Patient may have received prior treatment for their disease.
* Patient must have at least 3 months of follow-up from start of luspatercept treatment at the participating site.

Exclusion Criteria:

* Suspected or proven acute promyelocytic leukemia (APL) (FAB M3 or WHO 2008) based on morphology, immunophenotype, molecular assay or karyotype
* Currently enrolled in any interventional clinical trial where the patient is being treated with an investigational product that cannot be identified.
* Idiopathic Cytopenias of Undetermined Significance (ICUS), Myelodysplastic Syndromes (MDS) patients who received or are receiving active (disease modifying) therapy for the treatment of MDS prior to the date of informed consent.
* Acute Myeloid Leukemia (AML) patients who initiated active (disease modifying treatment for AML more than 2 weeks prior to the date of consent.
* Myelofibrosis (MF) and Myelodysplastic/Myeloproliferative (MDS/MPN) overlap syndrome patients with suspected juvenile myelomonocytic leukemia (JMML).

Luspatercept treated patients:

* Patient must not be currently or previously enrolled in the Connect Myeloid Registry.
* Patient must not have received luspatercept as part of a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Approximately 2,300 adult patients diagnosed with myeloid disease will be enrolled in Connect® Myeloid Registry from 200 sites (both community [70-80%] and academic [20-30%] facilities) across the US that are representative of where patients with myeloid diseases are diagnosed and treated.
Sampling Method: Non-Probability Sample
Enrollment: 2013 (Actual)
Dates: Start 2013-12-12 (Actual); Primary Completion 2024-10-18 (Actual); Study Completion 2024-10-18 (Actual)

PRIMARY OUTCOMES:
Patient Demographics- MDS/AML/ICUS Cohorts | Up to 8 years
  Describe demographics, baseline characteristics and clinical outcomes of the patients with LR or HR MDS, ICUS, and AML.
Diagnostic and Treatment Patterns- MDS/AML/ICUS Cohorts | Up to 8 years
  Describe current and evolving patterns for diagnosis, treatment sequencing, routine clinical practice patterns and clinical outcome measures in patients with LR or HR MDS, ICUS, and AML
Safety and Effectiveness- MDS/AML/ICUS Cohorts | Up to 8 years
  Describe the survival status, clinical response to treatment, select laboratory results, occurrence of secondary primary malignancies, deaths, select adverse events.
Patient Demographics- MF Cohort | Up to 5 years
  Describe demographics, baseline characteristics, patient recorded outcomes, and clinical outcomes of patients enrolled to the MF cohort
Diagnostic and Treatment Patterns- MF Cohort | Up to 5 years
  Describe current and evolving patterns for diagnosis, treatment sequencing, routine clinical practice patterns and clinical outcome measures in patients enrolled in the MF Cohort
Safety and Effectiveness- MF Cohort | Up to 5 years
  Describe the survival status, clinical response to treatment, select laboratory results, occurrence of secondary primary malignancies, deaths, select adverse events.
Treatment effectiveness - LTC | Minimum of 3-months post index date
  Describe clinical response to treatment, transfusion information, ECOG performance status and deaths.
Treatment patterns and clinical outcomes - LTC Cohort | Minimum of 3-months post index date
  Describe the myeloid malignancy treatment patterns and clinical outcomes before and after initiating luspatercept treatment
Transfusion information - LTC | Minimum of 3-months post index date
  Describe changes in hemoglobin and transfusion independence status.
Treatment duration - LTC Cohort | Minimum of 3-months post index date
  Luspatercept treatment duration

SECONDARY OUTCOMES:
Patient Reported Outcome | Up to 8 years
  Summarize patient reported outcomes (including e.g., Health-Related Quality of Life (HRQOL)) and economic outcomes, and their association with patient characteristics, treatment regimens, and clinical outcomes
Correlative Studies | Up to 8 years
  Perform molecular and cellular correlative studies on blood/bone marrow and oral epithelial cell samples.
Patient demographics and clinical characteristics - LTC | Baseline
  Describe demographics, baseline characteristics and clinical outcomes of the patients treated with luspatercept
Reason for treatment discontinuation - LTC | Minimum of 3-months post index date
  Describe reasons for luspatercept treatment discontinuation

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (157):
- United States (154):
  - DCH Health System (Lewis and Faye Manderson Cancer Center), Tuscaloosa, Alabama
  - Arizona Oncology, Phoenix, Arizona
  - The University of Arizona Cancer Center, Tucson, Arizona
  - Local Institution - 1273, Tucson, Arizona
  - Highlands Oncology Group, Fayetteville, Arkansas
  - Clopton Clinic of Jonesboro, Inc., Jonesboro, Arkansas
  - NEABC- Fowler Family Center for Cancer Care, Jonesboro, Arkansas
  - Local Institution - 1161, Jonesboro, Arkansas
  - Comprehensive Blood & Cancer Center, Bakersfield, California
  - Alta Bates Summit Comprehensive Cancer, Berkeley, California
  - Sutter East Bay Hospitals (dba Jordan Research and Education Institute - REDI), Berkeley, California
  - John Muir Clinical Research Center, Concord, California
  - VA Central California Health Care System, Fresno, California
  - UCSD Moores Cancer Center, La Jolla, California
  - Pacific Cancer Care, Monterey, California
  - Local Institution - 1016, San Diego, California
  - Local Institution - 1027, Santa Rosa, California
  - St. Joseph's Regional Cancer Center, Stockton, California
  - Saint Joseph Hospital, Cancer Centers of Colorado, Denver, Colorado
  - Regional Cancer Care Associates, Manchester, Connecticut
  - Bennett Cancer Center Stamford Hospital, Stamford, Connecticut
  - Delaware Clinical and Laboratory Physicians, Christiana, Delaware
  - University Cancer Institute, Boynton Beach, Florida
  - Halifax Health Center for Oncology, Daytona Beach, Florida
  - Holy Cross Hospital, Fort Lauderdale, Florida
  - University of Florida, Gainesville, Florida
  - Cancer Specialists of North Florida, Jacksonville, Florida
  - Watson Clinic Center for Cancer Care and Research, Lakeland, Florida
  - Ocala Oncology, Ocala, Florida
  - Adventist Health System/Sunbelt, Inc., Orlando, Florida
  - Memorial Healthcare System, Pembroke Pines, Florida
  - Sacred Heart Medical Oncology Group, Pensacola, Florida
  - Georgia Regents University Cancer Center, Augusta, Georgia
  - Southeast Georgia Health System, Brunswick, Georgia
  - Columbus Regional Research Institute, Columbus, Georgia
  - Northwest Georgia Oncology Centers, P.C., Marietta, Georgia
  - Saint Alphonsus Regional Medical Center, Boise, Idaho
  - RUSH University Cancer Center, Chicago, Illinois
  - NorthShore University Health System, Evanston, Illinois
  - Ingalls Memorial Hospital, Harvey, Illinois
  - Joliet Oncology Hematology Associates Ltd, Joliet, Illinois
  - Local Institution - 1145, Joliet, Illinois
  - Illinois Cancer Care, Peoria, Illinois
  - Quincy Medical Group, Quincy, Illinois
  - Edward H. KaPlan MD & Associates, Skokie, Illinois
  - Orchard Healthcare Research Inc., Skokie, Illinois
  - Simmons Cancer Institute at Southern Illinois University, Springfield, Illinois
  - St. Vincent Anderson Regional Hospital Research, Anderson, Indiana
  - IU health Bloomington Hospital, Bloomington, Indiana
  - Horizon Oncology Research, Inc, Lafayette, Indiana
  - McFarland Clinic, P.C, Ames, Iowa
  - Siouxland Hematology-Oncology Associates, Sioux City, Iowa
  - Central Care Cancer Center, Garden City, Kansas
  - Cotton O'Neil Clinical Research/ Stormont Vail Health, Topeka, Kansas
  - Cancer Center of Kansas, Wichita, Kansas
  - Mary Bird Perkins Cancer Center at St. Tammany, Covington, Louisiana
  - QCCA - Pontchartrain Cancer Center, Covington, Louisiana
  - Center for Cancer and Blood Disorders, Bethesda, Maryland
  - Maryland Oncology Hematology, Columbia, Maryland
  - Western Maryland Health System, Cumberland, Maryland
  - Carroll Regional Cancer Center, Westminster, Maryland
  - Cape Cod Hospital, Hyannis, Massachusetts
  - University of Michigan Health System (UMHS) - University Hospital (University of Michigan Medical Ce, Ann Arbor, Michigan
  - John D. Dingell VA Medical Center /Cynthia Marbury, Detroit, Michigan
  - Henry Ford Health System, Detroit, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Cancer and Hematology Centers of Western Michigan, Grand Rapids, Michigan
  - Ascension St. John Hospital_Hematology (was St. Johns Hospital and Hematology-Oncology Associates East PC ), Grosse Pointe Woods, Michigan
  - Michigan State University/Breslin Cancer Center, Lansing, Michigan
  - Essentia Health Oncology Clinical Trials, Duluth, Minnesota
  - Southdale Cancer Clinic, Edina, Minnesota
  - Metro MN CCOP/Park Nicollet Institute, Saint Louis Park, Minnesota
  - MCDA - Central Care Center, Bolivar, Missouri
  - Southeast Cancer Center, Cape Girardeau, Missouri
  - Boone Hospital Center, Columbia, Missouri
  - Harry S Truman Memorial Veterans' Hospital, Columbia, Missouri
  - Mercy Cancer Center - Joplin, Joplin, Missouri
  - Kansas City Veterans Affairs Medical Center, Kansas City, Missouri
  - Heartland Regional Medical Center (Heartland Health), Saint Joseph, Missouri
  - Mercy Research - Springfield, Springfield, Missouri
  - Local Institution - 1110, St Louis, Missouri
  - Missouri Baptist Medical Center, St Louis, Missouri
  - St. Vincent Frontier Cancer Center, Billings, Montana
  - Southeast Nebraska Cancer Center, Lincoln, Nebraska
  - VA Medical Center Manchester, Manchester, New Hampshire
  - John Theurer Cancer Center (Hackensack U Med Center), Hackensack, New Jersey
  - Saint Peter's University Hospital, New Brunswick, New Jersey
  - St Joseph Healthcare System, Paterson, New Jersey
  - Somerset Medical Center 110 Rehill Avenue, Somerville, New Jersey
  - Sparta Cancer Center, Sparta, New Jersey
  - Bassett Heathcare Network, Cooperstown, New York
  - Hematology Oncology Associates of Central NY, East Syracuse, New York
  - Huntington Medical Group, Huntington Station, New York
  - Local Institution - 1047, Johnson City, New York
  - Weill Cornell Medical College, New York, New York
  - Rochester General Hospital, Rochester, New York
  - St. Francis Hospital, Roslyn, New York
  - New York Cancer and Blood Specialists, The Bronx, New York
  - New York Medical College, Valhalla, New York
  - Leo W Jenkins Cancer Center, Greenville, North Carolina
  - Kinston Medical Specialists, Kinston, North Carolina
  - Summa Health System, Akron, Ohio
  - University Hospitals, Case Medical Center, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Local Institution - 1088, Cleveland, Ohio
  - Mid Ohio Oncology/Hematology, Inc., dba The Mark H. Zangmeister Center, Columbus, Ohio
  - University of Toledo Medical Center (Utmc), Toledo, Ohio
  - INTEGRIS Cancer Institute Southwest Medical Center, Oklahoma City, Oklahoma
  - INTEGRIS Cancer Institute of Oklahoma Proton Campus, Oklahoma City, Oklahoma
  - Oklahoma Cancer Specialist and Research Institute, Tulsa, Oklahoma
  - Local Institution - 1131, Portland, Oregon
  - Providence Cancer Center, Portland, Oregon
  - Salem Health, Salem, Oregon
  - Hematology and Oncology Assoc of NEPA, Dunmore, Pennsylvania
  - Lancaster Cancer Center, Lancaster, Pennsylvania
  - Lancaster General Hospital, Lancaster, Pennsylvania
  - Reading Hospital - McGlinn Cancer Institute, West Reading, Pennsylvania
  - Cancer Care Associates of York, York, Pennsylvania
  - Roger Williams Medical Center, Providence, Rhode Island
  - Prisma Health Cancer Institute - Upstate, Greenville, South Carolina
  - Spartanburg Regional Medical Center, Spartanburg, South Carolina
  - Prairie Lakes Health Systen, Inc, Watertown, South Dakota
  - Thompson Cancer Survival Center, Knoxville, Tennessee
  - University of Tennessee Medical Center Cancer Intitute, Knoxville, Tennessee
  - Regional One Health, Memphis, Tennessee
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee
  - Hendrick Cancer Center, Abilene, Texas
  - Texas Oncology, Amarillo Cancer Center, Amarillo, Texas
  - Dallas VA Medical Center, Dallas, Texas
  - HOLD - Texas Oncology, Dallas, Dallas, Texas
  - Texas Oncology - Sammons Cancer Center, Dallas, Texas
  - Oncology and Hematology of South Texas, PA, Laredo, Texas
  - Southwest Cancer Treatment & Research Center, Lubbock, Texas
  - Texas Oncology, McAllen (plus 2 satelite sites), McAllen, Texas
  - Scott & White Healthcare, Round Rock, Texas
  - Baylor Research Institute dba Scott & White Memorial Hospital, Temple, Texas
  - Community Cancer Trials of Utah, Ogden, Utah
  - VA Medical Center - White River Junction, White River Junction, Vermont
  - Lynchburg Hematology Oncology Clinic, Lynchburg, Virginia
  - Peninsula Cancer Institute, Newport News, Virginia
  - PeaceHealth St Joseph Cancer Center, Bellingham, Washington
  - Providence Regional Cancer Partnership, Everett, Washington
  - Kadlec Regional Medical Center (KRMC), Kennewick, Washington
  - Vista Oncology Inc. PS, Olympia, Washington
  - Benaroya Research Institute at Virginia Mason, Seattle, Washington
  - Swedish Cancer Institute, Seattle, Washington
  - Providence St. Mary Regional Cancer Center, Walla Walla, Washington
  - West Virginia University, Morgantown, West Virginia
  - St. Vincent Hospital, Green Bay, Wisconsin
  - Bellin Memorial Hospital/ Bellin Cancer Team, Green Bay, Wisconsin
  - Gundersen Lutheran Inc, La Crosse, Wisconsin
  - Columbia St. Mary'S, Milwaukee, Wisconsin
  - Wheaton Franciscan Cancer Care - All Saints, Racine, Wisconsin
  - Waukesha Memorial Hospital, Waukesha, Wisconsin
- Puerto Rico (3):
  - Puerto Rico Hematology Oncology Group, Bayamón
  - VA Caribbean Healthcare System CRADA, San Juan
  - Fundacion de lnvestigaci6n, San Juan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Steensma DP, Abedi M, Bejar R, Cogle CR, Foucar K, Garcia-Manero G, George TI, Grinblatt D, Komrokji R, Ma X, Maciejewski J, Pollyea DA, Savona MR, Scott B, Sekeres MA, Thompson MA, Swern AS, Nifenecker M, Sugrue MM, Erba H. Connect MDS/AML: design of the myelodysplastic syndromes and acute myeloid leukemia disease registry, a prospective observational cohort study. BMC Cancer. 2016 Aug 19;16:652. doi: 10.1186/s12885-016-2710-6. PMID 27538433
- [Derived] Patel JL, Erba HP, Savona MR, Grinblatt DL, Clark M, Clive TC, Smart TB, Makinde AY, DeGutis IS, Yu E, Eggington JM, George TI. Genomic Data Heterogeneity across Molecular Diagnostic Laboratories: A Real-World Connect Myeloid Disease Registry Perspective on Variabilities in Genomic Assay Methodology and Reporting. J Mol Diagn. 2023 Aug;25(8):611-618. doi: 10.1016/j.jmoldx.2023.05.002. PMID 37517825